CLINICAL TRIAL: NCT03839342
Title: Binimetinib and Encorafenib for the Treatment of Advanced Solid Tumors With Non-V600E BRAF Mutations
Acronym: BEAVER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEAVER-001 / IST-818-207X
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor
Keywords: Advanced Cancer; Advanced Solid Tumors; Non-V600 BRAF Mutations
MeSH Terms: interventions — binimetinib; encorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Binimetinib + Encorafenib (Experimental): Binimetinib and encorafenib are administered orally on a twice daily or once daily schedule, respectively in 28-day cycles. Treatment will continue until it is discontinued due to unacceptable toxicity, clinical or radiological disease progression as per RECIST 1.1, investigator decision, and/or withdrawal of consent.
  Interventions: Drug: Binimetinib; Drug: Encorafenib

INTERVENTIONS:
Drug: Binimetinib — MEK inhibitor, 45mg oral tablet
Drug: Encorafenib — BRAF inhibitor, 450mg oral capsule

SUMMARY:
This is a single-centre, open-label Phase II study of the investigational drugs binimetinib and encorafenib that will be taken my mouth (orally) daily in adult patient with advanced and/or metastatic solid tumors for which no other standard therapy is available. The main purpose is to evaluate the objective response rate (ORR) of the study drugs in the growth of the cancer in patients with class 2 and 3 BRAF mutations.

DETAILED DESCRIPTION:
BRAF is a gene in humans that is commonly altered in cancer, resulting in a change to the proteins created from this mutation. These altered proteins interact with a process in the body known as the MAPK (mitogen-activated protein kinase) pathway and promote the growth of cancer. Three classes of BRAF mutations have been identified to understand why some patients respond to treatment and others do not. Class 2 and 3 BRAF mutations have worse overall survival. This study will look at participants in these classes (non-V600E BRAF mutations).

Binimetinib is an oral drug (tablet) that stops the function of MEK (mitogen-activated protein kinase kinase). MEK is a part of the MAPK pathway, so blocking this step helps in stopping the pathway from confinuing to grow the cancer.

Encorafenib is an oral drug (capsule) that stops the function of BRAF V600-mutant kinase, the protein that is produced from a type of BRAF gene mutation. This protein promotes the MAPK pathway so blocking this protein stops the MAPK pathway from growing the cancer.

Patients will visit the clinic up to 2 times every 4 weeks (1 cycle) for tests and procedures while taking the study drugs daily. Procedures will involve review of medication and history, imaging scans, blood sample collection for safety and research purposes, urine collection, ECGs, eye exam, MUGA scans and mandatory and optional tumor biopsies.

ELIGIBILITY:
Inclusion Criteria:

Informed consent

1. Signed written and voluntary informed consent.
2. Patient must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
3. Age > 18 years, male or female.

   Disease characteristics
4. Patient must be diagnosed with a histologically or cytologically-documented, locally-advanced, or metastatic solid malignancy that is incurable and has either (a) failed prior standard therapy, (b) for which no standard therapy exists, or (c) standard therapy is not considered appropriate by the patient and treating physician.
5. Measurable disease by RECIST v1.1 criteria.
6. Malignancy must express one of the following BRAF alterations: BRAF mutation affecting codon: 241, 257, 367, 462, 463, 464, 466, 467, 469, 485, 581, 586, 594, 595, 596, 597 598, 599, 601; V600 BRAF mutations: V600K (for any malignancy except melanoma), V600D, V600M, V600R; BRAF deletions ie. V600_K601delinsE or 1799_1801 del TGA; BRAF insertions ie. T599dup; BRAF fusions ie. KIAA1549:BRAF
7. All patients enrolled must be willing and able to provide at least 1 archival and/or fresh tumor biopsy at baseline for histopathological and molecular evaluation during the screening period with binimetinib and encorafenib. Additional matched pre-treatment and on-treatment fresh tumor biopsies are mandatory for 10 patients enrolled in stage 2. Any patient with insufficient or inadequate archival tissue samples will be required to provide a fresh tumor biopsy. For all other patients, a fresh baseline biopsy is optional, but highly recommended. If a patient only has a single measurable lesion by RECIST v1.1, this lesion can be used for baseline biopsy if it is 2cm or greater.
8. Patient must be able to swallow pills
9. Patient must be willing to provide serial blood samples for molecular profiling of ctDNA evolution

   Patient characteristics
10. ECOG performance status 0-1.
11. Patient must have adequate organ function as determined by the following:

    • Renal function: i. Serum creatinine < 1.5 ULN (upper limit of normal range) or a calculated creatinine clearance of > 50mL/min using the following Cockcroft-Gault formula:

    Creatinine clearance = [(140-age) x wt (kg) x Constant*] / creatinine (umol/L)

    *Constant = 1.23 for men, and 1.04 for women

    • Bone marrow function (without hematopoietic growth factors or transfusion): i. Absolute neutrophil count (ANC) > 1.0 x 109/L ii. Leukocytes > 2.0 x 109/L iii. Hemoglobin > 90 g/L or > 9g/dL iv. Platelets > 75 x 109/L v. Previous blood transfusions are acceptable, however patients must have achieved the above hemoglobin and platelet targets without requiring a blood transfusion within 14 days prior to study entry.

    • Liver function: i. Total bilirubin ≤ 1.5 × ULN and < 35 uMol/L; OR total bilirubin >1.5 × ULN with indirect bilirubin < 1.5 × ULN. Total bilirubin < 1.5 x ULN or ≤ 3 x ULN for patients with Gilbert Syndrome.

    ii. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) < 2 x ULN, unless patients are known to have liver metastases. For patients with known liver metastases, Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) < 5 x ULN

    • Cardiac function: i. A normal left ventricular ejection fraction (LVEF) of ≥ 50% by a MUGA scan or echocardiogram performed within 4 weeks of the study commencement.

    ii. QTc interval ≤ 480 ms (triplicate ECGs)
12. Female participants of childbearing potential as described in Section 5.5.4, must have a negative serum β HCG test result.
13. Female participants of childbearing potential must agree to use methods of contraception that are highly effective or acceptable, as described in Section 5.5.4, and to not donate ova from Screening until 30 days after the last dose of study drug
14. Male participants must agree to use methods of contraception that are highly effective or acceptable, as described in Section 5.5.4, and to not donate sperm from Screening until 90 days after the last dose of study drug.
15. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

Patients meeting any of the following criteria are excluded from the study:

1. Any patient with a tumor expressing a BRAF V600E mutation
2. Any patient with melanoma whose tumor expresses a BRAF V600K mutation
3. Prior therapy with any BRAF inhibitor (e.g., encorafenib, dabrafenib, vemurafenib) and/or any MEK inhibitor (e.g., binimetinib, trametinib, cobimetinib).
4. Patients receiving any systemic chemotherapy, immunotherapy, or targeted therapy, within 4 weeks from the last dose prior to study treatment. The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment. Local treatment (e.g. by local surgery or radiotherapy) of isolated lesions for palliative intent is acceptable within 2 weeks, with prior consultation and in agreement with the principal investigator.
5. Any symptomatic brain metastasis Note: Patients previously treated or untreated for this condition who are asymptomatic in the absence of corticosteroid and anti-epileptic therapy are allowed. Brain metastases must be stable for ≥ 4 weeks, with imaging (e.g., magnetic resonance imaging [MRI] or computed tomography [CT]) demonstrating no current evidence of progressive brain metastases at screening.
6. History or current evidence of retinal vein occlusion (RVO) or current risk factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of retinal degenerative disease
7. Leptomeningeal disease
8. Previous or concurrent malignancy within 3 years of study entry, with the following exceptions: adequately treated basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, or other noninvasive or indolent malignancy; other solid tumors treated curatively without evidence of recurrence for at least 3 years prior to study entry (note: based on mechanism of action, BRAF inhibitors may cause progression of cancers associated with RAS mutations)
9. Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:
10. History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) <6 months prior to screening,
11. Symptomatic chronic heart failure (i.e. New York Heart Association Class ≥ 2), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality <6 months prior to screening except atrial fibrillation and paroxysmal supraventricular tachycardia;
12. Uncontrolled hypertension defined as persistent elevation of systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100mmHg, despite current therapy;
13. Known positive serology for HIV (Human immunodeficiency virus) that is not currently controlled with anti-retroviral therapy,
14. Has a known history of or is positive for active hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (defined as HCV RNA [qualitative] is detected). HBV DNA must be undetectable and HBsAg negative at Screening Visit. Participants who have had definitive treatment for HCV are permitted if HCV RNA is undetectable at Screening Visit.
15. Known history of acute or chronic pancreatitis. Patients with previous history of pancreatitis caused by immunotherapy are not excluded if pancreatitis is resolved.
16. History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) ≤ 12 months prior to starting study treatment
17. Impaired gastrointestinal function or disease that may significantly alter the absorption of encorafenib or binimetinib (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption)
18. History of known hypercoaguability risk factors (other than cancer) ie. Factor V Leiden. Patients with a history of previous DVT or PE who are currently asymptomatic and treated with anticoagulation therapy are allowed.
19. Concurrent neuromuscular disorder that is associated with the potential of elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
20. Patients who are planning on embarking on a new strenuous exercise regimen after first dose of study treatment. Note: Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on binimetinib treatment
21. Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., active infection/inflammation requiring systemic therapy, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc. Previous bacterial infections are acceptable if patients completed antibiotic course 3 days prior to initiating study treatment.
22. Patients who have undergone major surgery ≤ 3 weeks prior to starting study drug or who have not recovered from side effects of such procedure;
23. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test;
24. Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-06-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate defined as per RECIST v1.1. | 2.5 years

SECONDARY OUTCOMES:
Number of participants with toxicities as per NCI CTCAE v5.0. | 2.5 years
Disease progression defined as per RECIST v1.1 and monitored throughout the study period. Progression Free Survival defined as time from study registration to disease progression or death from any cause. | 2.5 years
Disease Control Rate defined in accordance with RECIST v1.1, as the percentage of patients who achieve a complete response, partial response or stable disease after 24 weeks of treatment. | 2.5 years
Overall survival measured as the length of time from the first day of treatment to the day of death. Median OS will be reported. | 2.5 years
Change in circulating tumor DNA (ctDNA) profiles measured by serial analysis of ctDNA profiles at baseline, mid-cycle 1, with each subsequent cycle, and at progression, validated by comparison to molecular profiles of corresponding fresh tumor biopsies | 2.5 years
Number of fresh tumor biopsies collected, frozen, and stored for subsequent development of patient derived xenografts. | 2.5 years
Number of identified molecular mechanisms of acquired resistance to binimetinib and encorafenib in tumors with non-V600E BRAF mutations, measured by analysis of molecular profiles and validated with PDX models in vitro and in vivo. | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna Spreafico, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Biomarker test results and limited clinical information that does not identify patients may be sent to centralized scientific databases or shared with collaborating researchers outside of UHN. Data from this study can be shared through two types of databases:
  Open-Access: publicly accessible and will contain limited clinical information and analyses of patient samples. It will not contain data that can identify an individual.
  Controlled-Access: will contain more detailed clinical information and sample analyses. It will be stripped of all personal identifiers. Researchers who use data from this database will sign agreements that define how data may be used. They will not be permitted to disclose or transfer data to others. They must use the data only for the approved purposes and must agree not to attempt to re-identify patients from their data.

REFERENCES:
- [Derived] Rajkumar S, Berry D, Heney KA, Strong C, Ramsay L, Lajoie M, Alkallas R, Nguyen TT, Thomson C, Ahanfeshar-Adams M, Dankner M, Petrella T, Rose AAN, Siegel PM, Watson IR. Melanomas with concurrent BRAF non-p.V600 and NF1 loss-of-function mutations are targetable by BRAF/MEK inhibitor combination therapy. Cell Rep. 2022 Apr 5;39(1):110634. doi: 10.1016/j.celrep.2022.110634. PMID 35385748